CLINICAL TRIAL: NCT05088746
Title: Comparing Different Timings for Periodontal Re-evaluation After Non-surgical Periodontal Therapy (NSPT)
Status: Recruiting | Type: Observational
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Prof Elena Calciolari, Principal Investigator. DDS, MS., PhD, University of Parma
Other Study IDs: P-002
Record Dates: First submitted 2021-05-27; First posted 2021-10-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis; Periodontal Pocket
MeSH Terms: conditions — Periodontitis; Periodontal Pocket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-stimulated saliva sample will be collected at certain visits (baseline, 3-4, 6-8 and 12 months post NSPT), and will be stored (frozen) for analysis.
  Samples of GCF will be collected from the deepest sites (maximum of 5) at baseline, 3-4, 6-8 and 12 months post NSPT. GCF will be collected prior to periodontal probing to avoid contamination by blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-surgical periodontal therapy
  Interventions: Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — NSPT will be performed following the principles of minimally invasive non-surgical therapy (MINST) described by Nibali et al. (Nibali et al., 2015, Nibali et al., 2019)

SUMMARY:
This is a prospective cohort study that aims to describe the difference in terms of percentage of closed pockets (PPD <5 mm and no BOP) when performing the periodontal re-evaluation at 3-4, 6-8 and 12 months.

Fifty-two, ≥18-year old, otherwise healthy, periodontitis patients will be recruited at Centro di Odontoiatria, Università di Parma.

DETAILED DESCRIPTION:
This is a prospective cohort study describing the difference in terms of percentage of closed pockets (PPD <5 mm and no BOP) when performing the periodontal re-evaluation at 3-4, 6-8 or 12 months. The trial will follow the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement. The study consists of 7 visits over a period of 15 months.

Visit 1 - Baseline -

* Informed consent, medical/dental history and demographics
* Record concomitant medications and smoking history
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, PI, mobility and furcation involvement. PPD, REC, PI and BOP will be recorded at 6 sites per tooth.
* Standardized peri-apical x-rays for the sites with PPD≥5mm, as per standard of practice (if not already available within the previous 6 months)
* Intra-oral 3D scan
* Oral hygiene instructions and demonstration of self-performed oral hygiene measures
* PROMs questionnaires
* Saliva collection and GCF collection from the deepest pockets (maximum of 5 sites)

Visit 2 and 3 - NSPT - (and extra visit 3.1 and 3.2 if needed) (within 60 days from baseline)

* Update medical/dental history and record adverse events and/or concomitant medications
* NSPT, consisting in the careful removal of hard and soft deposits with ultrasonic instruments at infected sites performed by an experienced clinician following the principles of minimally invasive non-surgical therapy (MINST). A quadrant approach will be adopted and it will be left to the discretion of the clinician to choose whether to instrument 1 or 2 quadrants at a time and the length of session visits. Hence, 2 to 4 sessions of NSPT with an interval of 1 week between each other will be performed. During NSPT, teeth considered hopeless will be extracted as per standard of practice.
* Reinforcement of oral hygiene instructions
* PROMs questionnaires

Extra visits outside the study protocol may be arranged in case the patients need extractions or other dental treatments besides NSPT.

Visit 4 (4-6 weeks from the end of NSPT)

* Update medical/dental history and record adverse events and/or concomitant medications
* Visual inspection of signs of inflammation and plaque
* Supragingival polish and reinforcement of oral hygiene instructions
* PROMs questionnaires
* Intra-oral 3D scan

Visit 5 (3-4 months from the end of NSPT)

* Update medical/dental history and record adverse events and/or concomitant medications
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, PI, mobility and furcation involvement. PPD, REC, PI and BOP will be recorded at 6 sites per tooth.
* PROMs questionnaires
* Intra-oral 3D scan
* Saliva collection and GCF collection from the same sites identified at baseline
* Supragingival polish and reinforcement of oral hygiene instructions

Visit 6 (6-8 months from the end of NSPT)

* Update medical/dental history and record adverse events and/or concomitant medications
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, PI, mobility and furcation involvement. PPD, REC, PI and BOP will be recorded at 6 sites per tooth.
* PROMs questionnaires
* Intra-oral 3D scan
* Saliva collection and GCF collection from the same sites identified at baseline
* Supragingival polish and reinforcement of oral hygiene instructions

Visit 7 (12 months ± 14 days from the end of NSPT)

* Update medical/dental history and record adverse events and/or concomitant medications
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, PI, mobility and furcation involvement. PPD, REC, PI and BOP will be recorded at 6 sites per tooth.
* PROMs questionnaires
* Intra-oral 3D scan
* Standardized peri-apical x-rays
* Saliva collection and GCF collection from the same sites identified at baseline
* Supragingival polish and reinforcement of oral hygiene instructions

Photos and videos may be taken/recorded in any of the study visits for documentation purposes. The subject will not be identifiable from those photos/videos.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy males and females ≥18 years old
* Willingness to read and sign a copy of the Informed Consent Form after reading the Patient Information Sheet, and after the nature of the study has been fully explained
* Clinical evidence of periodontitis, defined as the presence of interdental clinical attachment loss detectable at ≥2 non-adjacent teeth or buccal or oral clinical attachment loss ≥3mm with pocketing >3 mm detectable at ≥2 teeth (Tonetti et al., 2018)
* Not having received subgingival instrumentation within the previous 12 months

Exclusion Criteria:

* Medical history that includes serious medical conditions or transmittable diseases (e.g. serious cardiovascular disease, organ transplant, renal failure, AIDS, viral etc.).
* Antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam.
* In treatment with drugs that induce gingival overgrowth
* History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* History of alcohol or drug abuse.
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing, which can affect interpretation of study results).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in percentage of closed pockets (PPD <5 mm and no BOP) | From baseline to 3-4; 6-8 and 12 months

SECONDARY OUTCOMES:
Changes in probing pocket depth (PPD), recession (REC) and clinical attachment level (CAL) | From baseline to 3-4; 6-8 and 12 months
Changes in the percentages of sites with PPD reduction ≥2mm | From baseline to 3-4; 6-8 and 12 months
Changes in the percentages of sites with CAL gain ≥2mm | From baseline to 3-4; 6-8 and 12 months
Changes in the percentage of deep pockets (PPD≥6 mm) | From baseline to 3-4; 6-8 and 12 months
Evaluation of global changes in quality of life | 4-6 weeks; 3-4 months; 6-8 months; 12 months
  In all post NSPT re-evaluations (Visit 4 to 7), a questionnaire (2 questions) will be given to participants to assess changes in quality of life following periodontal therapy
changes in oral impact on daily performance (OIDP) | From baseline to 4-6 weeks; 3-4 months; 6-8 months; 12 months
  Self-administered questionnaire, it is a composite measure of the impacts of oral health on the quality of life of people.
Changes in global ratings of periodontal health and quality of life | From baseline to 4-6 weeks; 3-4 months; 6-8 months; 12 months
  self administered questionnaire and VAS scale
Evaluation of changes in patient perception about therapy | From non-surgical therapy visit to 4-6 weeks follow-up
  VAS scale to evaluate patient perception about therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitario di Odontoiatria, Parma, Italy

IPD SHARING:
Plan to Share IPD: No
Centro di Odontoiatria is the sponsor for this study. We will be using patient information in order to undertake this study and will act as the data controller for this study. This means that we are responsible for looking after patient information and using it properly. We will keep identifiable information for 20 years after the study has finished.
  The only people within the Centro di Odontoiatria who will have access to information that identifies the patients will be people who need to contact them about the research study, and make sure that relevant information about the study is recorded for their care, and to oversee the quality of the study or audit the data collection process. The people who analyse the information will not be able to identify patients and will not be able to find out their name or contact details.